CLINICAL TRIAL: NCT04471272
Title: Radiofrequency Ablation for Hepatocellular Carcinoma Using Gradual RF Energy Delivery Mode With Octopus Electrodes: A Prospective Observational Study
Brief Title: RFA Using Gradual RF Energy Delivery Mode With Octopus Electrodes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-1909-086-1064
Record Dates: First submitted 2020-03-31; First posted 2020-07-15 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Radiofrequency Ablation; Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: * Study population: RFA using gradual RF energy delivery mode with Octopus electrodes
  * Control group: Over a period of two years from 2017 to 2018, the patients who performed RFA for HCC using octopus electrodes and the maximum high-frequency energy transfer mode technique were collected. After performing propensity score matching analysis using variables of liver function values, the same number of controls are selected and set.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RFA using gradual RF energy delivery mode (Experimental): RFA therapy is performed on HCC less than 4 cm in size using an octopus electrode, a double-shift unipolar high-frequency transmission mode, and a gradual high-frequency energy loading mode.
  Interventions: Procedure: RFA using gradual RF energy delivery mode with Octopus electrodes

INTERVENTIONS:
Procedure: RFA using gradual RF energy delivery mode with Octopus electrodes — RFA therapy is performed on HCC less than 4 cm in size using an octopus electrode, a double-shift unipolar high-frequency transmission mode, and a gradual high-frequency energy loading mode.

SUMMARY:
The investigators intend to perform RFA therapy on HCC less than 4 cm in size using octopus electrode, double alternating unipolar high-frequency transmission mode and gradual high-frequency energy loading mode, and to find out the therapeutic results. The primary evaluation variable is the ideal technical success rate for securing a safety margin of 5 mm or more around the tumor on the CT obtained immediately after the procedure, and the secondary evaluation variable is the volume of the cauterization lesion per unit time measured on the CT obtained immediately after the procedure, The local tumor recurrence rate, survival rate and disease-free survival rate of 12 months after the procedure, the presence or absence of multiple recurrences within the same segment, the actual procedure time, and the incidence of complications associated with the procedure are examined. The performance of RFA therapy of HCC using the Octopus electrode and gradual high-frequency energy transfer mode is compared with that of the existing Octopus electrode and RFA therapy using the basic maximum high-frequency energy transfer mode using historic cohort.

DETAILED DESCRIPTION:
1. Pre-treatment planning:

   The detailed plan of radio frequency ablation (RFA) will be implemented in accordance with the routine procedure of image evaluation prior to high frequency implementation. In other words, the location of the tumor on the Multiphasic CT or MRI and the RFA planning program at the 3D workstation (Philips, Intraportal) before RFA procedure, evaluate the tumor volume and the relationship with adjacent blood vessels, and insert the electrode for RFA After planning the number of ablation and the like, the location of the tumor in the ultrasound image was found in the pre-surgery image by fusion of the pre-surgery image and the ultrasound image using US-CT-MR fusion and contrast-enhanced ultrasonography, which are recently used. It will evaluate whether the tumors match, and also evaluate whether the distribution of the echo bubble and the tumor position coincide during the procedure in real time.

   In addition, the degree of stiffness of the parenchyma will be measured by using an ultrasound elastic technique. At this time, the ultrasonic fusion device to be used will be one of Phillips, GE, or one of the navigation systems of Siemens, Canon, and Samsung, available here. The fused image guides the location of the electrodes to be installed in the tumor, the number of electrodes, and a safe access route. If the extent of the tumor is not clearly visible, or the image before the procedure is too old (> 6 weeks), low kVp or DECT will be conducted to evaluate the tumor's extent more accurately.
2. RFA procedure As the equipment of RFA, the multi-VIVA generator and octopus electrode used herein will be used. In the method of treatment, three high-frequency electrode needles were placed on the tumor according to the clinical need under the guidance of fusion ultrasound, and then the electrodes were cooled with saline, and the two electrodes were simultaneously applied with high-frequency waves for approximately 6-30 minutes depending on the size of the tumor. The temperature is maintained at 90-100 degrees Celsius. At this time, the high-frequency energy is increased by 10W at 30W intervals at 60Watt for the first 3 minutes, and then gradually increased by 10W per minute after 100W.

The location of the tumor on the ultrasound image by fusion of the ultrasound image with the pre-procedure using the US-CT-MR fusion tool (Navigator- GE, PercuNav-Phillips, Canon, S-fusion: Samsung), which is frequently used in RFA procedures. It will evaluate whether the tumors found in the images before the procedure match, and also evaluate whether the distribution of the echo bubble and the tumor location coincide during the procedure in real time. At this time, the navigation systems used by Samsung, Phillips, GE, and Canon will be used as the ultrasonic fusion device to be used. In the Fusion US image, the Octopus electrode is safely placed in the tumor through the access path of the electrode already planned. Thereafter, while transmitting high-frequency energy, air bubbles are generated in the tumor on the ultrasound image, and an echogenic cloud is formed while the procedure is stopped when the echogenic cloud becomes larger than 5 mm than the tumor.

ELIGIBILITY:
Inclusion Criteria:

* agree to the protocol's requirements and submit a consent form
* 20 years old-85 years old
* Child-Pugh Class A
* among patients with chronic hepatitis or cirrhosis, MDCT or MRI hepatocellular carcinoma of less than 4 cm in size was suspected, and was referred to the radiology department considering clinical RFA therapy as a clinical judgment.

Exclusion Criteria:

* when the number of malignant HCC is 3 or more
* if the tumor has a maximum size of more than 4 cm
* diffuse infiltrative HCC
* Child-Pugh class B or C
* If there is an invasion of liver vessels due to malignant HCC
* severe coagulopathy
* multiple distant metastasis
* situations where it is very unlikely to obtain appropriate data for research purposes

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Ideal technical success rate | Time: immediately
  Secure a safety margin of 5 mm or more around the tumor on CT obtained immediately after the procedure

SECONDARY OUTCOMES:
Ablation volume | Time: immediately
  Volume of ablation lesions per unit time measured on CT obtained immediately after the procedure
Local recurrence rate | Time: 12months
  Local recurrence rate of 12 months after the procedure
Overall survival rate | Time: 3years
  Survival rate after the procedure
Disease free survival | Time: 3years
  disease-free survival rate after the procedure
Complication rate | Time: immediately
  The incidence of complications associated with the procedure
Technical time | Time: immediately
  The actual procedure time

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No